CLINICAL TRIAL: NCT04122027
Title: Use of Cerebral Oximetry In Adult Chinese Patients For Liver Transplantation
Brief Title: A Prospective Randomized Controlled Trial on the Use of Cerebral Oximetry in Adult Chinese Patients Undergoing Liver Transplantation
Acronym: LT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kenneth Siu-Ho Chok, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UW 18-321
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Patients undergoing liver transplantation without regional cerebral oxygenation monitoring using a cerebral oximeter.
  Interventions: Other: Cerebral oximeter
- Intervention (Active Comparator): Patients undergoing liver transplantation with regional cerebral oxygenation monitoring using a cerebral oximeter.
  Interventions: Other: Cerebral oximeter

INTERVENTIONS:
Other: Cerebral oximeter — Near infra-red spectroscopy, NIRS

SUMMARY:
Liver transplantation (LT) is a life-saving procedure for patients with end-stage liver diseases. Although with continuous advancement in technology, it remains a high-risk operation. The goal of LT is not only ensure survival of the patients but also to restore them back to their pre-morbid state with a good quality of life. Neurological sequelae can have major impact on postoperative outcomes after LT and yet the reported literature is scarce. Studies from Western countries showed some evidence on the use of cerebral oximtery in cardiac surgery to prevent neurological mishaps. LT shares similar intra-operative fluctuation of the haemodynamices as in cardiac surgery, causing disturbances in regional cerebral oxygenation and theorectically cerebral oximetry should be of great value as well in LT surgery. Data from a large randomised controlled trial is lacking from the current literatures. We therefore propose a prospective randomized controlled trial on the use of this device in adult LT and see whether its use could reduce neurological mishaps.

DETAILED DESCRIPTION:
Liver Transplant Liver transplantation (LT) is a life-saving procedure for patients with end-stage liver disease. Despite continuous advancement in technology, it remains a high-risk operation. The building-up of an oxygen debt during LT can lead to an increased risk of poor postoperative outcomes (1, 2). Furthermore, patients with acute liver failure or end-stage liver disease are prone to hepatic encephalopathy, which can lead to disturbance of auto-regulation in the brain, which may eventually cause cerebral hypoxia and ischaemia. Irresversible metabolic disturbances can impair cerebral auto-regulation, causing poor neurological outcomes after LT (3). The prevalence of encephalopathy, delirium and stroke in transplant recipients is 12-40% (3). Hypotheses for these conditions include prolonged stay in the intensive care unit (ICU) (so-called "ICU psychosis"), the use of Tacrolimus (4), rapid correction of hyponatraemia (5) and impaired cerebral auto-regulation (3), but no definite conclusion can be made most of the time. Among these hypotheses, impairment of cerebral auto-regulation has never been documented in large clinical trials for Chinese patients in LT.

Cerebral oximetry (Near infra-red spectroscopy, NIRS) There is no "gold standard" for measuring cerebral auto-regulation. Monitoring of the brain oxygenation, such as direct tissue O2 tension and jugular bulb O2 saturation, has been used as a surrogate of auto-regulation but it is invasive. Transcranial laser Doppler (TCD) of the middle cerebral artery has been validated in healthy volunteers as well as real patients as a good measurement of cerebral blood flow (6, 7). Similarly, near-infrared spectroscopy (NIRS), a non-invasive and continuous method, can also monitor the regional cerebral oxygenation (rScO2) and is increasingly used in cardiac surgery. A previous report has validated the use of NIRS when compared to TCD, as the latter requires a trained technician to monitor and supervise. NIRS provides a timely, real-time, inexpensive, easily measurable alternative to TCD, and thus should have a great potential for clinical usage in LT. Similar to other non-invasive oximetry (e.g. pulse oximetry), measurement can be done through adhesive tapes over bilateral forehead and connected to the machine (INVOS™ 5100C Cerebral/Somatic Oximeter by Covidien). This system is the ONLY cerebral/somatic oximetry system with FDA cleared improved outcome claims (8). Plachky et al. showed that 50% of patients demonstrated a decline in cerebral oxygen saturation when clamping of the vessles during LT and it had positive correlation with the postoperative cerebral disrubances (9). Nonetheless, the clinical application for patients undergoing LT is scarce and its application is novel. The use of this technology may potenitally be limited by the presence of high levels of bilirubin acting as a chromophore interferring with its data acquistion. However, in a pilot study of 9 patients who underwent LT investigators using this technology were able to demonstrate that 3 out of 9 patients had either transient or persistent impaired auto regulation throughout the operation. This in turn was associated with higher Model of End-Stage Disease Score (MELD) >15 (p=0.015), more postoperative seizures and stroke (P<0.0001) (3). A recent systematic review (10) of 901 Caucasians from 24 publications showing a decrease in NIRS (>15% relative to baseline) could have impaired postoperative cognitive function (28 versus 26; MMSE) and reduced LOS (14 versus 23 days) in open surgery. In the field of LT, impaired cerebral autoregulation (25%), cerebral deoxygenation in the anhepatic phase (36%) and cerebral hyperoxygenation with reperfusion of the grafted liver (14%) were identified by NIRS and could lead to adverse neurological outcome such as seizures, transient hemiparesis and stroke. Nonetheless, no large prospective randomized trial and no Chinese cohort were included.

References

1. Shoemaker WC, Appel PL, Kram HB. Role of oxygen debt in the development of organ failure sepsis, and death in high-risk surgical patients. Chest. 1992;102(1):208-15.
2. Shoemaker WC, Appel PL, Kram HB. Hemodynamic and oxygen transport responses in survivors and nonsurvivors of high-risk surgery. Critical care medicine. 1993;21(7):977-90.
3. Lescot T, Karvellas CJ, Chaudhury P, Tchervenkov J, Paraskevas S, Barkun J, et al. Postoperative delirium in the intensive care unit predicts worse outcomes in liver transplant recipients. Can J Gastroenterol. 2013;27(4):207-12.
4. DiMartini AF, Trzepacz PT, Pajer KA, Faett D, Fung J. Neuropsychiatric side effects of FK506 vs. cyclosporine A. First-week postoperative findings. Psychosomatics. 1997;38(6):565-9.
5. Lee J, Kim DK, Lee JW, Oh KH, Oh YK, Na KY, et al. Rapid Correction Rate of Hyponatremia as an Independent Risk Factor for Neurological Complication Following Liver Transplantation. Tohoku J Exp Med. 2013;229(2):97-105.
6. Lang EW, Mehdorn HM, Dorsch NW, Czosnyka M. Continuous monitoring of cerebrovascular autoregulation: a validation study. Journal of neurology, neurosurgery, and psychiatry. 2002;72(5):583-6.
7. Ono M, Zheng Y, Joshi B, Sigl JC, Hogue CW. Validation of a stand-alone near-infrared spectroscopy system for monitoring cerebral autoregulation during cardiac surgery. Anesthesia and analgesia. 2013;116(1):198-204.
8. Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, et al. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesthesia and analgesia. 2007;104(1):51-8.
9. Plachky J, Hofer S, Volkmann M, Martin E, Bardenheuer HJ, Weigand MA. Regional cerebral oxygen saturation is a sensitive marker of cerebral hypoperfusion during orthotopic liver transplantation. Anesth Analg. 2004;99(2):344-9.
10. Sorensen H, Grocott HP, Secher NH. Near infrared spectroscopy for frontal lobe oxygenation during non-vascular abdominal surgery. Clin Physiol Funct Imaging. 2016;36(6):427-35.

ELIGIBILITY:
Inclusion Criteria:

* Able to get informed consent by patient
* Patients undergo DDLT or LDLT at Department of Surgery, Liver Transplant Centre, The University of Hong Kong, Queen Mary Hospital
* Ethnicity is Chinese

Exclusion Criteria:

* Refusal of consent by patient
* Pre-existing neurological damage, history of seizures and on antidepressants
* Skin conditions over forehead that precludes the application of sensors of equipment
* Ethnicity is not Chinese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Duration of confusion as assessed by the Confusion Assessment method | 48 hours after liver transplant
  To assess patients experience of development of delirium

SECONDARY OUTCOMES:
The time taken for MOCA to return to baseline | 10 days after liver transplant
  To assess the time patients required to return health conditions within 10 days after surgery
Other complications unrelated to neurological deficit according to Clavien-Dino Classification. | 2 years
  To monitor any other complications developed by patients after liver transplant

CONTACTS AND LOCATIONS:
Locations (2):
- Queen Mary Hospital, Hong Kong, China
- Queen mary Hospital, Hong Kong, Hong Kong